CLINICAL TRIAL: NCT06302023
Title: Docosahexaenoic Acid (DHA) Supplementation During Pregnancy Reduces the Risk of Preterm Birth in Threatened Preterm Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Wiphawi Phattharachindanuwong, Fellow, Maternal and Fetal medicine department, Obstetrics and gynecology department, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE661462
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Pregnant Women Diagnosed With Threatened Preterm Labor
Keywords: DHA; threatened preterm labor; Docosahexaenoic acid
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA supplement (Experimental): DHA supplement 1000mg per day
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA) 1000 mg
- no DHA supplement (No Intervention): no DHA supplement

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) 1000 mg — Pregnant women will be ask to take a DHA 1000 mg per days at bedtime until delivery or 37 week of gestational age
  Other Names: NOW
  Arms: DHA supplement

SUMMARY:
The goal of this clinical trial is to learn about the effects of Docosahexaenoic acid (DHA) in reducing the incidence of premature birth in threatened preterm labor

The main questions it aims to answer are:

* Can DHA supplementation reduce the incidence of premature birth in threatened preterm labor?
* How does DHA supplementation affect pregnancy outcomes? Participants were organized into two groups
* Group 1 (Intervention) Participants will be asked to take a DHA 1000mg per day
* Group 2 (control) Participant will not need to take a DHA

DETAILED DESCRIPTION:
Threatened preterm labor is defined as regular uterine contractions occurring before 37 completed weeks of gestation, without any cervical dilation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Between 24 wk to 34 wk of gestational age
* Pregnant women diagnosed threatened preterm labor (with no cervical change)

Exclusion Criteria:

* Fetal anomalies
* Multiple pregnancy
* Premature rupture of membrane
* Placental disorders: placenta previa, placental abruption
* Fetal growth restriction
* Pregnancy complication: gestational diabetes mellitus, Chronic hypertension
* Allergic reaction to DHA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with preterm birth | at delivery time
  Delivery at less than 37 weeks of gestational age

SECONDARY OUTCOMES:
Rate of low birth weight neonate | at delivery time
  Newborn's weight at birth is less than 2500g
Rate of Neonatal Intensive care unit admission | at delivery time
  newborn need neonatal intensive care

CONTACTS AND LOCATIONS:
Locations (1):
- KhonKaenU, Khon Kaen, KhonKaen, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year 4 months

REFERENCES:
- [Derived] Phattharachindanuwong W, Chaiyarach S, Komwilaisak R, Saksiriwuttho P, Duangkum C, Kongwattanakul K, Kleebkaow P, Waidee T, Pongsamakthai M, Chantanavilai S, Srisataporn T. Docosahexaenoic acid (DHA) Supplementation During Pregnancy Reduces the Risk of Preterm Birth in Threatened Preterm Labor. The Multicenter Randomized Controlled Trial. Int J Womens Health. 2025 Mar 30;17:937-945. doi: 10.2147/IJWH.S518312. eCollection 2025. PMID 40183030